CLINICAL TRIAL: NCT01640145
Title: Impact of Acute Low Intensity Exercise and Protein Intake on Skeletal Muscle Protein Synthesis in Elderly: a Randomized Controlled Trial
Brief Title: Effect of Low Intensity Exercise and Protein Intake on Skeletal Muscle Protein Synthesis in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Jakob Agergaard, MSc, PhD Student, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BBH98
Record Dates: First submitted 2012-07-09; First posted 2012-07-13 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Skeletal Muscle Protein Synthesis in Elderly; Protein Kinetics; Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Proteins; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Carbohydrate (Placebo Comparator)
  Interventions: Other: Exercise
- Protein continous boluses (Active Comparator)
  Interventions: Dietary Supplement: Protein; Other: Exercise
- Protein 2 boluses (Active Comparator)
  Interventions: Dietary Supplement: Protein; Other: Exercise

INTERVENTIONS:
Dietary Supplement: Protein — Whey protein intake
  Arms: Protein 2 boluses; Protein continous boluses
Other: Exercise — Unilateral low intensity exercise

SUMMARY:
Maintenance of skeletal muscle mass is crucial during lifespan to retain health and functional autonomy. Sarcopenia, being the loss of muscle mass during aging, is a well-known phenomenon in the elderly and a major challenge viewed from an individual, and a socioeconomic point of view. Nevertheless, several studies have proved muscle tissue to be markedly affected by physical activity and nutritional interventions even at old age. Recently, a study in young individuals showed that an acute bout of easily tolerated low intensity exercise can prolong the muscle building effects of a milk protein intake compared to a non-exercised situation. Therefore, the major aim of the present project is to evaluate, whether a low intensity exercise regime in conjunction with milk protein supplementation can induce positive adaptations on parameters related to muscle size and function in elderly.

The study focuses on the acute muscle protein synthesis response to low intensity exercise and protein supplementation measured with stable isotope tracer techniques. It is hypothesized that light muscle activity can augment and prolong the effects of protein feeding.

If a light resistance exercise protocol as investigated in the present project can prove beneficial, elderly, frail elderly, and individuals undergoing rehabilitation can challenge sarcopenia in a new and tolerable way.

ELIGIBILITY:
Inclusion Criteria:

* Male
* >65 year old
* Healthy
* BMI <28

Exclusion Criteria:

* Smoker
* Type II diabetic
* Intake of medicine or supplements which will affect skeletal muscle protein synthesis
* Alcohol intake >21 units/week.
* Frequent exercise or hard physical labor

Min Age: 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-07; Primary Completion 2013-01 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle protein synthesis | 6 months
  Measured as myofibrillar fractional synthetic rate (%/hour) in three periods pre intervention: 0-3 hours, 3-7 hours and 7-10 hours

SECONDARY OUTCOMES:
Gene expression | 1.5 years
  Through real time RT-PCR we measure the fold changes in gene expression of targets involved in skeletal muscle remodeling: myogenic factors, atrogenes, matrix related genes
Intracellular signaling | 1.5 years
  Through Western Blotting we will measure changes in intracellular hypertrophy signaling. That is the activity of protein targets from the Akt-mTORC1 and Akt-FOXO pathways.
Amino acid transporter | 2 years
  Through Western Blotting and RT-PCR protein and mRNA expression of amino acid transporters (LAT1, SNAT2, PAT1) are analyzed

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sports Medicine Copenhagen, Copenhagen, Copenhagen, Denmark